CLINICAL TRIAL: NCT02096562
Title: Prospective Randomized Assessment of Postsurgical Swelling Applying Compression Stockings vs. Conventional Wrapping After Outpatient Surgery
Brief Title: Knee Swelling Under Use of Compression Stockings After Outpatient Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rostock (Other)
Responsible Party: Principal Investigator, Sebastian Oye, University of Rostock, University of Rostock
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A 2013-0083
Record Dates: First submitted 2013-11-11; First posted 2014-03-26 (Estimated); Last update posted 2016-05-24 (Estimated); Status verified 2016-05

CONDITIONS: Knee Pain Swelling
Keywords: knee welling outpatient compression stockings
MeSH Terms: interventions — Postoperative Period

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- B - No compression stockings (Placebo Comparator): normal therapy - no compression stockings
  Interventions: Other: normal therapy - no compression stockings
- A - Use of compression stockings (Active Comparator): Patients use compression stockings for 10 days after surgery
  Interventions: Other: Patients use compression stockings for 10 days after surgery

INTERVENTIONS:
Other: Patients use compression stockings for 10 days after surgery — patients wear compression stocking for 24 hours in the first 2 days after surgery and for at least 8 hours at day 3-10 after surgery
  Arms: A - Use of compression stockings
Other: normal therapy - no compression stockings — the patients receive the common therapy according to S2 guidelines
  Arms: B - No compression stockings

SUMMARY:
Outpatients who undergo knee surgery are designated two different clinical study groups. Group A receives common wrapping after surgery to the first postsurgical day and will be provided with compression stockings for the following 10 days, while group B only receives common wrapping and will not be provided with compression stockings.

The investigators are going to investigate the effect of compression stockings on postsurgical swelling and formation of edema on outpatients.

DETAILED DESCRIPTION:
The investigators are planing on investigate the effect of compression stockings on postsurgical swelling and formation of edema. For this purpose the investigators devide outpatients who have undergone knee surgery to two different clinical study groups. Group A receives a common compression bandage after surgery to the first postsurgical day and receives compression stockings afterwards for the following 10 days, while Group B only receives a common compression bandage to the first postsurgical day. Group A will be instructed to wear compression stockings for 24 hours on the first two postsurgical day, afterwards at least for 8 hours a day.

Preoperatively the investigators are going to determine the volume and circumference of both legs using the Bodytronic 600 by Bauerfeind. Subsequently the measurement will be repeated on the first, forth and tenth postsurgical day. The investigators are going to measure the range of motion, also the patients of both groups will be asked to mark pain and tension on a visual analog scale and write down the amount of time they have been lying, sitting and standing each day. Group A will document the amount of time for how long they were wearing compression stockings each day.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years
* signed release form

Exclusion Criteria:

* deep vein thrombosis
* swelling caused by cardiac, venous or endocrine genesis
* dysfunction of the lymphatic system
* dysfunction of kidney or liver
* Use of water withholding medication
* massive adiposity
* cachexia
* epilepsy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2013-07; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Amount of Swelling of lower Extremity (circumference in mm and volume in ml) | 10 days

SECONDARY OUTCOMES:
Pain (visual analoge scale) and Range of Movement (degree of flexion) | 10 days

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Tischer, Prof. Dr., Study Director — OUK Rostock
Locations (1):
- Orthopädische Klinik und Poliklinik - Universitätsmedizin Rostock, Rostock, Meckenburg-Vorpommern, Germany

REFERENCES:
- [Derived] Tischer TS, Oye S, Lenz R, Kreuz P, Mittelmeier W, Bader R, Tischer T. Impact of compression stockings on leg swelling after arthroscopy - a prospective randomised pilot study. BMC Musculoskelet Disord. 2019 Apr 9;20(1):161. doi: 10.1186/s12891-019-2540-1. PMID 30967135